CLINICAL TRIAL: NCT05683691
Title: Prospective, Multicenter, Single-Arm Study of VanquishTM Water Vapor Ablation for PrOstate CanceR
Brief Title: Water Vapor Ablation for Localized Intermediate Risk Prostate Cancer
Acronym: VAPOR 2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Francis Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4760-001
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, Multicenter, Single-Arm Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Vanquish System Treatment (Experimental)
  Interventions: Device: Vanquish System

INTERVENTIONS:
Device: Vanquish System — Water vapor ablation delivered transurethrally in patients with intermediate risk, localized prostate cancer.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Vanquish Water Vapor Ablation Device ("Vanquish") in treating subjects with Gleason Grade Group 2 (GGG2) localized intermediate-risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. ≥50 years of age; with life expectancy of ≥10 years
2. 20-80 cc prostate size determined by MRI Central Imaging
3. ≤15 ng/ml PSA
4. Cancer stage less than or equal to T2c
5. Within 12 months prior to signing consent have had a multiparametric MRI. Within 6 months prior to signing consent, have undergone a multiparametric MRI software guided fusion biopsy of the prostate (transrectal or transperineal). This must include a standard sector biopsy obtaining a minimum of 10 cores.

   * <15mm diameter of qualifying lesion as measure by greatest diameter
6. Subject is willing and able to adhere to specific protocol visits and required testing throughout study
7. Is geographically stable and near the site or able and willing to travel back to site for follow-up visits involving diagnostic tests or treatment
8. Able and willing to provide written consent to participate in the study.
9. Subject is willing and able to be treated within 180 days after signing consent.

Exclusion Criteria:

1. Patients with >GGG3 cores anywhere in the prostate
2. MRI evidence of extracapsular extension of cancer (MRI read as "definite", "frank" or "gross" ECE)
3. All MRI Central Imaging confirmed PI-RADS 5 lesions
4. All MRI Central Imaging confirmed additional PI-RADS 4 lesions.
5. Contraindications to MRI
6. Subjects with an installed pacemaker or other potentially electrically conductive implants implanted within 200mm (8 inches) of the procedure area. Implants that are within 200mm (8 inches) and can be turned off for the duration of the study procedure are acceptable.
7. Any prior surgery, intervention, or minimally invasive therapy, (MIST) for the prostate cancer or bladder neck.
8. Treated within the past 5 years for genital cancer
9. Presence of any urethral or prostatic condition that precludes water vapor ablation per Instructions for Use
10. Currently taking medications that have hormonal effects on the prostate or PSA, such as: 5 alpha reductase inhibitors (if on for <6 months, 6-month washout), Androgen blockers, Luteinizing hormone-releasing hormone (LHRH) agonists or antagonists (12-month washout), or Testosterone supplementation (3-month washout)
11. Active urinary tract infection. Subjects with an active infection who can be treated and re-tested with a negative result within the screening window are acceptable.
12. Active or clinically chronic prostatitis or granulomatous prostatitis
13. Treated within the past 5 years for a lower and/or upper urinary tract malignancy.
14. Any previous treatment for prostate cancer.
15. Any rectal pathology, anomaly or previous treatment that could change properties of rectal wall or insertion and use of TRUS
16. Unable to stop taking antiplatelet medications or other blood thinning agents
17. Known allergy to nickel
18. Allergic to medication required by the study such as MRI contrast or anesthesia
19. Any significant medical history that would pose an unreasonable risk or make the subject unsuitable for the study
20. Any cognitive or psychiatric condition that interferes with or precludes direct and accurate communication with the study Investigator regarding the study or affects the ability to complete the study quality of life questionnaires
21. Subject currently participating in other premarket investigational studies unless approved by Sponsor in writing
22. Subject is considered vulnerable such as incarcerated or cognitively impaired.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 36 months
  Freedom from systemic disease AND systemic therapy AND salvage therapy AND GGG≥2.
Primary Safety Endpoint | 12 months
  The proportion of subjects free from new or worsening urinary incontinence based on pad use at 12 months will be statistically compared to a performance goal.

SECONDARY OUTCOMES:
Key Secondary Endpoint | 36 months
  The proportion of subjects free from impotence.

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Mayo Clinic- Phoenix, Phoenix, Arizona
  - Memorial Care, Laguna Hills, California
  - University of Southern California, Los Angeles, California
  - Kasraeian Urology, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - Wichita Urology, Wichita, Kansas
  - WK Advanced Urology Specialists, Shreveport, Louisiana
  - Chesapeake Urology, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Corewell Health / William Beaumont University Hospital, Royal Oak, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic- Rochester, Rochester, Minnesota
  - Minnesota Urology, Woodbury, Minnesota
  - NYU Langone Health, New York, New York
  - Northwell Health- Lenox Hill Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Duke Cancer Institute, Durham, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Austin, Austin, Texas
  - Houston Methodist Hospital and Research Institute, Houston, Texas
  - The Urology Place, San Antonio, Texas
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No